CLINICAL TRIAL: NCT00592631
Title: Assessment of the Effects of Short and Long Term Use of Continuous Positive Airway Pressure on Airway Reactivity in Children and Adults With and Without Asthma
Brief Title: Assessment Of The Effects Of Short and Long Term Use Of CPAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Key investigator resigned
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0405-16; 0405-16
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Results first posted 2016-02-10 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-01

CONDITIONS: Asthma
Keywords: asthma; sleep apnea
MeSH Terms: conditions — Asthma; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP (Experimental): Subjects will use CPAP of 8-12 during days 2 through 6 of the study.
  Interventions: Device: CPAP-Continuous Positive Airway Pressure
- SHAM (Sham Comparator): Subjects will use sham CPAP of 0-2 during days 2 through 6 of the study.
  Interventions: Device: SHAM

INTERVENTIONS:
Device: CPAP-Continuous Positive Airway Pressure — Cpap will be worn at night by subjects 6 to 7 days duration.
  Arms: CPAP
Device: SHAM — SHAM will be worn at night by subjects 6 to 7 days duration.
  Arms: SHAM

SUMMARY:
We hypothesize that the nocturnal use of continuous positive airway pressure in adults and children with asthma will decrease airway reactivity.

DETAILED DESCRIPTION:
Deep inspirations have been shown to decrease the sensitivity of airways to narrowing (airway reactivity) after inhalation of agents that induce constriction of the bronchi in healthy adults. This response is absent in adult asthmatics; however, there is data demonstrating that use of continuous positive airway pressure (CPAP) for short periods of time may decrease airway reactivity in adult asthmatics. This suggests that although deep inspirations may not result in decreased airway reactivity, sustained lung inflation may lead to changes in asthmatic airway smooth muscle structure that lead to a decrease in airway reactivity. The purpose of our study is to determine whether short and long term use of CPAP in children and adults leads to decreased airway reactivity. If airway reactivity is decreased with CPAP, this may provide a novel therapeutic strategy for patients with asthma.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for children 8-18

* Children 8-18 years of age scheduled to start CPAP for obstructive sleep apnea.
* Subjects can have clinically stable asthma, with no plans by their physician to change asthma therapy over the next month

Inclusion criteria adults 18-60

* Adults 18-60 years of age, seen in adult Pulmonary Clinic for sleep related problems who may require treatment with nocturnal continuous positive pressure (CPAP), which will be determined by polysomnography(PSG) will be approached to participate in the study.

Exclusion Criteria:

Exclusions for Children category age 8-18 include:

1. Cyanotic congenital heart disease.
2. History of acute respiratory symptoms for 3 weeks prior to testing.
3. Inability to perform pulmonary function testing adequately.
4. Escalation in asthma medication at time of recruitment.
5. SaO2 <93% while awake and breathing room air
6. Baseline FEV1 <75% predicted

Exclusions for adults 18-60 include:

1. Gastro-Esophageal Reflux requiring Medical management.
2. Chronic Obstructive Pulmonary Disease.
3. Use of Supplemental Oxygen.
4. Ischemic Heart Disease or Hypertension requiring treatment with medications other than diuretics.
5. Use of systemic corticosteroid therapy during the past 6 months.
6. Acute Respiratory Illness in the previous 8 weeks.

Exclusions/Inclusion criteria for adults with asthma include:

1. Juniper Score <1.5
2. Baseline FEV1 > or equal to 70%
3. Non-smoking for 6 months
4. Less than 10 pack year smoking history
5. No change in asthma medications for the last 2 months
6. Negative pregnancy test
7. Subject cannot have sleep apnea

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2005-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. Tepper, MD, PhD, Principal Investigator — Indiana University; Mike Busk, MD, Study Director — NIFS/ Indiana University
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Busk M, Busk N, Puntenney P, Hutchins J, Yu Z, Gunst SJ, Tepper RS. Use of continuous positive airway pressure reduces airway reactivity in adults with asthma. Eur Respir J. 2013 Feb;41(2):317-22. doi: 10.1183/09031936.00059712. Epub 2012 Jul 26. PMID 22835615

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous Positivie Airway Pressure: Adult with stable asthma and normal spirometry used CPAP with a mask pressure between 8 and 10 cm H20 for 7 to 10 nights prior to the follow-up assessment.
- Sham Treatment: Adults with stable asthma and normal spirometry used SHAM with a mask pressure Mask pressure between 0 and 2 cm H20 for 7 to 10 nights prior to the follow-up assessment.
Period: Overall Study
Arm/Group | Continuous Positivie Airway Pressure | Sham Treatment
Started | 16 | 11
Completed | 16 | 9
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- CPAP: Subjects used CPAP set at 8-10 cmH20 for 7-10 nights.
- Sham: Subjects used SHAM set at 0-2 cmH20 for 7-10 nights
- Total: Total of all reporting groups
Arm/Group | CPAP | Sham | Total
Number analyzed (Participants) | 16 | 9 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (6) | 32 (9) | 29 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Provocative Concentration of Methacholine Causing a 20% Fall in Forced Expiratory Volume in 1 Second (FEV1)
Description: Methacholine is an inhaled medication used to assess asthma and reactive airways. It was given at increasing concentrations (beginning with 0.0625 mg/ml and ending with 16.0 mg/ml). Each dose was followed by a lung measurement until a change of FEV1 of 20% occurs or until a maximum dose was reached, whichever came first.
Time Frame: 7 to 10 nights after cpap is started.
Measure: Mean (Standard Error); unit: log mg/ml
Arm/Group | CPAP | Sham
Number analyzed (Participants) | 16 | 9
log mg/ml | 0.406 (0.066) | 0.003 (0.193)

ADVERSE EVENTS:
Arm/Group | Continuous Positive Airway Pressure | Sham
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/9
Other Adverse Events (participants affected / at risk) | 0/16 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No